CLINICAL TRIAL: NCT01911819
Title: A Histomorphometric Analysis of Bone Formation With Three Different Bone Graft Materials Following Sinus Augmentation
Brief Title: A Comparison of Bone Formation With Three Different Bone Graft Materials Following Sinus Graft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Collaborators: American Regent, Inc. (Industry)
Responsible Party: Principal Investigator, Joseph Kan, DDS, Professor of Restorative Dentistry, Loma Linda University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 5130213
Record Dates: First submitted 2013-07-18; First posted 2013-07-30 (Estimated); Results first posted 2017-12-13 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-11

CONDITIONS: Inadequate Bone Height in Maxillary Posterior Area
Keywords: Histomorphometric Analysis; New bone Formation; Sinus Augmentation; Bone Graft Materials
MeSH Terms: interventions — Sinus Floor Augmentation; equimatrix; Bio-Oss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sinus augmentation using Bio-oss (Experimental): Sinus augmentation using Bio-oss
  Interventions: Procedure: Sinus augmentation; Drug: Bio-oss
- Sinus augmentation using Equimatrix (Experimental): Sinus augmentation using Equimatrix
  Interventions: Procedure: Sinus augmentation; Drug: Equimatrix
- Sinus augmentation using OSSIF-i sem (Experimental): Sinus augmentation using OSSIF-i sem
  Interventions: Procedure: Sinus augmentation; Drug: OSSIF-i sem

INTERVENTIONS:
Procedure: Sinus augmentation
Drug: Equimatrix — Equimatrix cancellous particle size 0.2-1mm approximately 2g (4cc)
  Arms: Sinus augmentation using Equimatrix
Drug: OSSIF-i sem — OSSIF-i sem Mineralized Cancellous Bone Allograft SP 0.25-1.0mm approximately 2cc x 2
  Arms: Sinus augmentation using OSSIF-i sem
Drug: Bio-oss — Bio-oss small granules cancellous 0.25-1mm, approximately 2g (4cc)
  Arms: Sinus augmentation using Bio-oss

SUMMARY:
The purpose of this study is to compare new bone formation following bone graft in sinus using three different commercially available bone graft materials. The study hypothesis is that there is no difference in new bone formation among three bone graft materials under microscope.

DETAILED DESCRIPTION:
The purpose of this investigation is to compare new bone formation through histomorphometric analysis following maxillary sinus augmentation using three different bone graft materials. Null Hypothesis is that there is no histomorphometric difference in new bone formation in maxillary sinuses augmented using three different materials; anorganic bovine bone graft (Bio-Oss), anorganic equine bone graft (Equimatrix) and mineralized bone allograft (OSSIF-i sem). Patients who require sinus augmentation prior to implant placement will be selected to participate in this study. All patients will be randomly placed into three groups according to bone graft materials that will be used. Group A (Control group,n=10): Maxillary sinus augmentation using anorganic bovine bone graft (Bio-Oss), Group B (Test group,n=10):Maxillary sinus augmentation using anorganic equine bone graft (Equimatrix), and Group C (Test group,n=10):Maxillary sinus augmentation using mineralized bone allograft (OSSIF-i sem). All the patients will be treated with the same surgical technique consisting of sinus floor augmentation via a lateral approach.After a full-thickness flap reflection to expose the lateral wall of the sinus each antrostomy will be outlined with a carbide round bur and sinus membranes will be carefully elevated. If a perforation to the sinus membrane occurs, and if the perforation is < 5 mm in diameter and is able to be repaired, the surgeon will continue the procedure. Any perforation > 5 mm will be excluded from this study. Bone graft materials will be placed into the each sinus compartment for the three groups. After 8 months of healing, biopsy specimen will be collected from the previous antrostomy sites. Histomorphometric measurements of the percentage of vital bone of the area of bone. The percentage of non-bone material (allograft or xenograft) and the percentage of connective tissue will be also analyzed. Then the primary hypothesis will be analyzed statistically.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years old who are able to read and sign written consent form.
2. Patient who has good oral hygiene (Full-mouth plaque score <25%).
3. Subject would be available for study monitoring.
4. Patients with missing teeth in the maxillary posterior region who will require sinus augmentation f or implant placement. The patients may be partially or completely edentulous.
5. Delayed implant placement approximately 8 months following sinus grafting.

Exclusion Criteria:

A medical history that will complicate the outcome of the study such as:

1. alcohol, drug dependency,
2. signs or symptoms of maxillary sinus disease,
3. current smoker,
4. history of head and neck radiation treatment,
5. poor health or any other medical, physical or psychological reason that might affect the surgical procedure or the subsequent prosthodontic treatment and/or required follow-up examinations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-12; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Kan, DDS, MS, Principal Investigator — Loma Linda University School of Dentistry
Locations (1):
- Loma Linda University School of Dentistry, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The enrolled patients had either unilateral or bilateral maxillary sinus requiring maxillary sinus graft. For patients with bilateral sinus, each maxillary sinus was randomly assigned different treatment groups.
Units Other Than Participants: Maxillary Sinuses
Groups:
- Sinus Augmentation Using Equimatrix: Sinus augmentation using Equimatrix
  Sinus augmentation
  Equimatrix: Equimatrix cancellous particle size 0.2-1mm approximately 2.5g (5cc)
- Sinus Augmentation Using Bio-oss: Sinus augmentation using Bio-oss
  Sinus augmentation
  Bio-oss: Bio-oss small granules cancellous 0.25-1mm, approximately 2.5g (5cc)
- Sinus Augmentation Using OSSIF-i Sem: Sinus augmentation using OSSIF-i sem
  Sinus augmentation
  OSSIF-i sem: OSSIF-i sem Mineralized Cancellous Bone Allograft SP 0.25-1.0mm approximately 5cc
Period: Overall Study
Arm/Group | Sinus Augmentation Using Equimatrix | Sinus Augmentation Using Bio-oss | Sinus Augmentation Using OSSIF-i Sem
Started | 10; 10 Maxillary Sinuses | 11; 11 Maxillary Sinuses (One of 10 sinuses was replaced to another sinus due to infection.) | 10; 10 Maxillary Sinuses
Completed | 9; 9 Maxillary Sinuses | 9; 9 Maxillary Sinuses | 10; 10 Maxillary Sinuses
Not Completed | 1; 1 Maxillary Sinuses | 2; 2 Maxillary Sinuses | 0; 0 Maxillary Sinuses
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Either partially or completely edentulous posterior maxilla were included. In event of a bilateral maxillary sinuses, each maxillary sinus was randomly assigned different groups. Therefore, the number of participants overlaps. Two sinuses in Bio-Oss group, 1 sinus in Equimatrix group were removed from the study according to the study protocol.
Units Other Than Participants: Maxillary sinus
Groups:
- Total: Total of all reporting groups
Arm/Group | Sinus Augmentation Using Bio-oss | Sinus Augmentation Using Equimatrix | Sinus Augmentation Using OSSIF-i Sem | Total
Number analyzed (Participants) | 9 | 9 | 10 | 21
Number analyzed (Maxillary sinus) | 9 | 9 | 10 | 28
Age, Continuous [Mean (Full Range); unit: years] — Population: The numbers of analyzed were based on the numbers of maxillary sinuses, therefore, the total number of unique participants is different.
  years | 60.9 [33 to 75] | 65.6 [54 to 72] | 57.9 [29 to 75] | 61.5 [29 to 75]
Age, Customized [Number; unit: participants]
  Between 18 and 65 years | 5 | 4 | 6 | 11
  >=65 years | 4 | 5 | 4 | 10
Sex/Gender, Customized [Number; unit: participants]
  Female | 5 | 3 | 5 | 11
  Male | 4 | 6 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Vital Bone in a Total Amount of a Bone Specimen
Description: Bone biopsy was taken in a mean of 9.1 months after sinus graft procedure from previous lateral window of maxillary sinus. The bone cores were analyzed though histomorphometric analysis.
Time Frame: 24months
Measure: Mean (Standard Deviation); unit: percentage of vital bone
Units Other Than Participants: Maxillary sinuses
Arm/Group | Sinus Augmentation Using Bio-oss | Sinus Augmentation Using Equimatrix | Sinus Augmentation Using OSSIF-i Sem
Number analyzed (Participants) | 9 | 9 | 10
Number analyzed (Maxillary sinuses) | 9 | 9 | 10
percentage of vital bone | 10.9 (8.9) | 9.1 (5.9) | 32.0 (12.4)

2. Secondary Outcome: The Percentage of Non-vital Bone/Residual Bone Graft Material in a Bone.
Description: as for outcome 1
Time Frame: 24months
Measure: Mean (Standard Deviation); unit: percentage of residual bone materials
Units Other Than Participants: Maxillary Sinuses
Arm/Group | Sinus Augmentation Using Bio-oss | Sinus Augmentation Using Equimatrix | Sinus Augmentation Using OSSIF-i Sem
Number analyzed (Participants) | 9 | 9 | 10
Number analyzed (Maxillary Sinuses) | 9 | 9 | 10
percentage of residual bone materials | 34.3 (12.1) | 38.9 (5.3) | 5.5 (5.7)

ADVERSE EVENTS:
Time Frame: Adverse event was monitored up to 2 weeks.
Arm/Group | Sinus Augmentation Using Bio-oss | Sinus Augmentation Using Equimatrix | Sinus Augmentation Using OSSIF-i Sem
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 1/11 | 0/10 | 0/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sinus Augmentation Using Bio-oss (N=11) | Sinus Augmentation Using Equimatrix (N=10) | Sinus Augmentation Using OSSIF-i Sem (N=10)
Maxillary sinus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — An acute sinus infection was noted in one sinus in the group of sinus augmentation using Bio-Oss. The graft materials were removed. maxillary sinus compartment was cleaned, irrigated and the area was sutured after the sinus graft procedure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No